CLINICAL TRIAL: NCT04705818
Title: Combining Epigenetic And Immune Therapy to Beat Cancer. CAIRE Study
Brief Title: Combining Epigenetic And Immune Therapy to Beat Cancer.
Acronym: CAIRE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: AstraZeneca (Industry); Epizyme, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB2019-04; 2019-003303-35 (EudraCT Number)
Record Dates: First submitted 2021-01-11; First posted 2021-01-12 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumor; Advanced Colorectal Carcinoma; Advanced Soft-tissue Sarcoma; Advanced Pancreatic Adenocarcinoma; Adult Solid Tumor
Keywords: tertiary lymphoid structure; pancreatic cancer; soft-tissue sarcoma; immunotherapy; colorectal cancer; solid tumor; epigenetic
MeSH Terms: conditions — Tertiary Lymphoid Structures; Pancreatic Neoplasms; Sarcoma; Colorectal Neoplasms | interventions — durvalumab; tazemetostat

STUDY DESIGN:
Intervention Model Description: 4 independant single-arm, phase II trials, based on 2-stage Simon's optimal design:
  * cohort A: pancreatic cancer
  * cohort B: not MSI-H or MMR-deficient colorectal cancer
  * cohort C: metastatic solid tumor with positive interferon gamma signature and/or prensece of tertiary lymphoid structure
  * cohort D: soft-tissue sarcoma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort A: pancreatic cancer (Experimental): Patients with pancreatic cancer will be treated by durvalumab prescribed in association with tazemetostat
  Interventions: Drug: Durvalumab; Drug: Tazemetostat
- Cohort B: not MSI-H or MMR-deficient colorectal cancer (Experimental): Patients with colorectal cancer will be treated bydurvalumab prescribed in association with tazemetostat
  Interventions: Drug: Durvalumab; Drug: Tazemetostat
- Cohort C: metastatic solid tumor (Experimental): Patients with metastatic solid with positive interferon gamma signature and/or presence of tertiary lymphoid structurestumor will be treated bydurvalumab prescribed in association with tazemetostat
  Interventions: Drug: Durvalumab; Drug: Tazemetostat
- Cohort D: soft-tissue sarcoma (Experimental): Patients with soft-tissue sarcoma will be treated by durvalumab prescribed in association with tazemetostat
  Interventions: Drug: Durvalumab; Drug: Tazemetostat

INTERVENTIONS:
Drug: Durvalumab — Durvalumab will be administered by intraveinous infusion (1120 mg) on day 1, every 3 weeks. Treatment by durvalumab will start on Day 22 (i.e., day 1 of cycle 2)
Drug: Tazemetostat — Tazemetostat will be administered per-os, twice daily (800 mg x 2), continuously. Treatment by tazemetostat will start on day 1 (of cycle1).

SUMMARY:
Umbrella study structure to independently and simultaneously assess the effects of the association of durvalumab and tazemetostat in multiple solid tumors.

DETAILED DESCRIPTION:
4 independant, multicenter, prospective, signle-arm phase II trials, based on 2-stage Simon's optimal design, will be conducted in parallel to assess the efficacy of durvalumab when prescribed with tazemetostat, separately, in distinct cohorts of solid tumors:

* cohort A: patients with pancreatic cancer
* cohort B: patients with colorectal cancer not MSI-H or MMR-deficient
* cohort C: patients with metastatic solid tumors with positive interferon gamma signature and/or tertiary lymphoid structure positive
* cohort D: patients with soft-tissue sarcoma

ELIGIBILITY:
Inclusion Criteria:

1. Histology: histologically confirmed solid tumors including pancreatic cancer (cohort A), non MSI-H or MMR-deficient colorectal cancer (cohort B), solid tumor with positive IFNG gene expression signature and/or tertiary lymphoid structure positive (cohort C), soft-tissue sarcomas (Cohort D). Other solid tumor types may be included through future amendment of the current version of the study protocol.

   Note: for cohort C, IFNG gene expression and/or presence of tertiary lymphoid structure will be centrally assessed. Cohort D, diagnosis must be confirmed and reviewed by the RRePS Network.as recommended by the French NCI (Inca).
2. For cohort C, availability of archived FFPE tumor tissue sample for IFNG gene expression assessment and/or determination of the presence of tertiary lymphoid structure,
3. Advanced disease defined as metastatic or unresectable locally advanced disease,
4. Age ≥ 18 years,
5. ECOG, Performance status ≤ 1,
6. Measurable disease according to RECIST
7. Life expectancy > 3 months,
8. Participant must have advanced disease and must not be a candidate for other approved therapeutic regimen known to provide significant clinical benefit based on investigator judgment,
9. Adequate hematological, renal, metabolic and hepatic functions
10. No prior or concurrent malignant disease diagnosed or treated in the last 2 years except for adequately treated in situ carcinoma of the cervix, basal or squamous skin cell carcinoma, or in situ transitional bladder cell carcinoma,
11. At least three weeks since last chemotherapy, immunotherapy or any other pharmacological treatment and/or radiotherapy,
12. Recovery to grade ≤ 1 from any adverse event (AE) derived from previous treatment, excluding alopecia of any grade and non-painful peripheral neuropathy grade ≤ 2
13. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to inclusion.
14. Both women and men must agree to use a highly effective method of contraception throughout the treatment period and for at least nine months after discontinuation of treatment for women and six months after discontinuation of treatment for men.
15. Voluntary signed and dated written informed consents prior to any specific study procedure,
16. Participants with a social security in compliance with the French law.

Exclusion Criteria:

1. Previous treatment with durvalumab or tazemetostat,
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or CTLA-4 antibody,
3. EGFR/ALK/ROS mutated NSCLC,
4. Evidence of progressive or symptomatic central nervous system or leptomeningeal metastases,
5. Participation to a study involving a medical or therapeutic intervention in the last 30 days,
6. Previous enrolment in the present study,
7. Participant unable to follow and comply with the study procedures because of any geographical, familial, social or psychological reasons,
8. Known hypersensitivity to any involved study drug or of its formulation components,
9. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent
10. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 14 days prior to the first dose of trial treatment,
11. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia, or evidence of active pneumonitis on screening chest CT scan or interstitial lung disease with ongoing signs and symptoms at inclusion. History of radiation pneumonitis in the radiation field (fibrosis) is permitted,
12. Has known active tuberculosis, hepatitis B or hepatitis C,
13. Has a known history of Human Immunodeficiency Virus or known acquired immunodeficiency syndrome,
14. Persistent proteinuria > 3.5 g/24 hours measured by urine protein-creatinine ratio from a random urine sample (≥ Grade 3, NCI-CTCAE v5),
15. Major surgical procedure or significant traumatic injury within 28 days before inclusion,
16. Non-healing wound, non-healing ulcer, or non-healing bone fracture,
17. Participants with evidence or history of any bleeding diathesis, irrespective of severity,
18. Any hemorrhage or bleeding event ≥ CTCAE Grade 3 within 4 weeks prior to inclusion,
19. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 months before inclusion (except for adequately treated catheter-related venous thrombosis occurring more than one month before inclusion),
20. Ongoing infection > Grade 2 as per NCI CTCAE v5,
21. Uncontrolled hypertension (Systolic blood pressure > 140 mmHg or diastolic pressure > 90 mmHg) despite optimal medical management,
22. Congestive heart failure ≥ New York Heart Association class 2,
23. Unstable angina, new-onset angina (begun within the last 3 months),
24. Myocardial infarction less than 6 months before inclusion,
25. Uncontrolled cardiac arrhythmias,
26. Pregnant or breast-feeding participants,
27. Individuals deprived of liberty or placed under legal guardianship,
28. Prior organ transplantation, including allogeneic stem cell transplantation,
29. Known alcohol or drug abuse,
30. Participants with any condition that impairs their ability to swallow and retain tablets,
31. Other severe acute or chronic medical conditions including immune inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study,
32. Participant with anti-Vitamine K oral anticoagulation therapy,
33. Suspected or known intraabdominal fistula,
34. Screening QTc interval > 480 msec is excluded,
35. Has received a live vaccine within 30 days prior to the first dose of trial treatment.
36. Participants with a prior history of myeloid malignancies, including myelodysplastic syndromes (MDS), acute myeloid leukemia (AML) or myeloproliferative neoplasm (MPN),
37. Participants with a prior history of T-cell lymphoblastic lymphoma (T-LBL) / T-cell lymphoblastic leukemia (T-ALL).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Estimated)
Dates: Start 2021-07-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of antitumor activity of durvalumab combined with tazemetostat for cohort A | Within 6 months of treatment onset
  Antitumor activity will be assessed in terms of disease control rate, defined as complete response (CR), partial response (PR) and stable disease (SD) as per RECIST v1.1 criteria
Assessment of antitumor activity of durvalumab combined with tazemetostat for cohort B | Within 6 months of treatment onset
  Antitumor activity will be assessed in terms of disease control rate, defined as CR, PR and SD as per RECIST v1.1 criteria
Assessment of antitumor activity of durvalumab combined with tazemetostat for cohort C | Within 6 months of treatment onset
  Antitumor activity will be assessed in terms of objective response rate, defined as CR and PR as per RECIST v1.1 criteria
Assessment of antitumor activity of durvalumab combined with tazemetostat for cohort D | 6 months
  Antitumor activity will be assessed in terms of 6-months progression-free rate, defined as CR, PR and SD as per RECIST v1.1 criteria

SECONDARY OUTCOMES:
Assessment of antitumor activity of durvalumab combined with tazemetostat for cohort D | Within 6 months of treatment onset
  Antitumor activity will be assessed in terms of objective response rate, defined as CR and PR as per RECIST v1.1 criteria
Assessment of antitumor activity of durvalumab combined with tazemetostat for cohort A | 6 months
  Antitumor activity will be assessed in terms of 6-months progression-free rate, defined as CR, PR and SD as per RECIST v1.1 criteria
Assessment of antitumor activity of durvalumab combined with tazemetostat for cohort B | 6 months
  Antitumor activity will be assessed in terms of 6-months progression-free rate, defined as CR, PR and SD as per RECIST v1.1 criteria
Assessment of antitumor activity of durvalumab combined with tazemetostat for cohort C | 6 months
  Antitumor activity will be assessed in terms of 6-months progression-free rate, defined as CR, PR and SD as per RECIST v1.1 criteria
6-month objective response (OR) independently for each population | 6 months
  Objective response is defined as the proportion of patients with complete response (CR) or partial response (PR) observed at 6 months, based on RECIST 1.1 criteria
Best overall response, independently for each population | Throughout the treatment period, an expected average of 6 months
  Best overall response is defined as the best response across all time points (RECIST 1.1). The best overall response is determinded once all the data for the patient is known (RECIST 1.1)
1-year progression-free survival, independently for each population | 1 year
  Progression-free survival is defined as the delay between the start date of treatment and the date of progression (as per RECIST 1.1) or death (from any cause), whichever occurs first
1-year overall survival, independently for each population | 1 year
  Overall survival is defined as the delay between the start date of treatment and the date of death (of any cause)
Safety profile, independently for each population: Common Terminology Criteria for adverse events version 5 | Throughout the treatment period, an expected average of 6 months
  Toxicity graded using the Common Terminology Criteria for Adverse Events vers 5
Tumor immune cell levels | before treatment onset, cycle 2 day 1 and cycle 3 day 1 (each cycle is 21 days)
  Levels of immune cells in tumors will be measured by immunohistochemistry
Blood cytokines level | before treatment onset, cycle 2 day 1, cycle 3 day 1 and treatment discontinuation (each cycle is 21 days)
  Levels of cytokines in blood will be measured by ELISA
Blood lymphocytes level | before treatment onset, cycle 2 day 1, cycle 3 day 1 and treatment discontinuation (each cycle is 21 days)
  Levels of lymphocytes in blood will be measured by flow cytometry
Blood kynurenin level | before treatment onset, cycle 2 day 1, cycle 3 day 1 and treatment discontinuation (each cycle is 21 days)
  Levels of kynurenin in blood will be measured by ELISA

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Institut Bergonie, Bordeaux
  - CHRU Brest, Brest
  - CHU Poitiers, Poitiers

IPD SHARING:
Plan to Share IPD: No